CLINICAL TRIAL: NCT02997774
Title: Evaluation of the Effects of Cooler Dialysate on Liver Perfusion, Endotoxemia and Uremic Toxin Handling in Hemodialysis Patients
Brief Title: Cooler Dialysis and Liver Perfusion and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chris McIntyre (Other)
Responsible Party: Sponsor-Investigator, Chris McIntyre, Professor of Medicine, UWO, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 108616
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Haemodialysis Complication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Neither subjects nor the investigator at the study visits will be blinded; however, analysis of imaging data will be performed with the operator blinded to allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Dialysis (Active Comparator): Patient will undergo dialysis at 36.5 degrees Celsius to assess if this affects the liver function and perfusion
  Interventions: Other: Standard Dialysis
- Cooler Dialysis (Experimental): Patient will undergo dialysis at 35 degrees Celsius to assess if this affects the liver function and perfusion
  Interventions: Other: Cooler dialysis

INTERVENTIONS:
Other: Cooler dialysis — Having dialysis at a slightly cooler temperature (35 vs 36.5 degrees Celsius)
  Arms: Cooler Dialysis
Other: Standard Dialysis — Having dialysis at a standard temperature (36.5 degrees Celsius)
  Arms: Standard Dialysis

SUMMARY:
Having hemodialysis affects the blood supply to various organs in the body including the heart and the brain. With time, these effects build up and can affect the way these organs function. The investigators have previously shown that the liver (a key organ which works to help clean the blood, make proteins and turn all your food into energy) is also affected. One of the ways to help protect organs from injury due to dialysis has been cooling during dialysis. The investigators want to examine whether cooling during dialysis protects the blood supply to the liver. CT imaging will be used to measure this blood supply during hemodialysis with standard and cooler settings.

DETAILED DESCRIPTION:
Hemodialysis exerts significant hemodynamic effects with widespread consequences on vulnerable vascular beds. Cardiac injury, including myocardial stunning and subclinical myocardial ischemia, appears to be common and associated with significantly increased mortality. The liver has been shown to have preserved blood flow due to its dual blood supply. Even so, the liver excretory function is decreased and endotoxin levels in the blood increase during hemodialysis. Extracorporeal cooling during dialysis has been associated with protective effects on the brain and heart of dialysis patients. The effects of cooler dialysis on liver perfusion, function and endotoxemia during hemodialysis is unknown.

The investigators therefore propose to use CT perfusion imaging to examine the effect of cooling during hemodialysis on liver perfusion, relating this effect to endotoxin translocation and myocardial dysfunction. Additionally, they intend to investigate the potential effects on hepatic function in this context, examining the relationship between liver perfusion and endotoxemia, the metabolism of uremic toxins and clinical symptoms of uremia.

This is a prospective randomized cross-over study involving a single center recruiting patients from the prevalent dialysis population of London Health Sciences Centre (LHSC) Renal Program. Once recruited, patients will undergo two study hemodialysis sessions - one will use standard dialysate temperature of 36.5 degrees Celsius (HD36.5) and one will use cooler dialysate temperature at 35 degrees Celsius (HD35). The order of these two sessions will be randomly allocated. Before, during and after each session, participants will undergo cardiac and hepatic assessment. This will include CT scans, 2D echocardiography and indocyanine green (ICG) clearance measurements. In addition, participants will answer a number of questionnaires about uremic symptoms and blood tests will also be done.

The investigators' aim is to characterize and compare liver function and perfusion before during and after hemodialysis, with standard and cooler dialysate temperature.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide informed consent
* Age greater than 18 years
* Hemodialysis for at least 3 months
* No significant residual renal function (<250mls urine/day)

Exclusion Criteria:

* Chronic liver disease of any stage
* Chronic intestinal disease excluding Irritable Bowel Syndrome (IBS)
* Previous liver transplant or liver resection
* Previous Transjugular Portosystemic Shunt (TIPSS) insertion
* Active infection or malignancy
* Pregnant, breastfeeding or intending pregnancy
* Unable to give consent or understand written information
* Diabetic and experiencing hypoglycemia during dialysis within the last 2 months
* Known allergy/intolerance to contrast agent or iodides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Change in regional liver perfusion in mls/min/100g from baseline to peak stress during dialysis (3 hours into the dialysis session) with standard versus cooler dialysate temperature. | 2 years

SECONDARY OUTCOMES:
Change in global liver perfusion in mls/min/100g pre, during and post-dialysis with cooler dialysate | 2 years
ICG clearance rate pre, during and post-dialysis with cooler vs standard dialysate | 2 years
Contribution of portal venous flow to hepatic perfusion (PV fraction) pre, during and post-dialysis with cooler vs standard dialysate | 2 years
Endotoxin levels with cooler vs standard dialysate | 2 years
Troponin T levels with cooler vs standard dialysate | 2 years
Number of stunned myocardial segments with cooler vs standard dialysate | 2 years
Uremic toxin levels with cooler vs standard dialysate | 2 years
Uremic symptom scores with cooler vs standard dialysate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chris W McIntyre, PhD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No